CLINICAL TRIAL: NCT01249105
Title: A Phase II Study of MK-2206 for Recurrent Malignant Glioma
Brief Title: MK-2206 for Recurrent Malignant Glioma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Merck (supplier of study drug & funding) has undergone a large reprioritization, in which they had to terminate many oncology trials, including this one.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Memorial Sloan Kettering Cancer Center (Other); University of California, Los Angeles (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Patrick Y. Wen, MD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-160; 018-00 (Other: Merck)
Record Dates: First submitted 2010-11-24; First posted 2010-11-29 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Malignant Glioma
Keywords: MK-2206; GBM
MeSH Terms: conditions — Glioma | interventions — MK 2206

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part 1 (Experimental): Patients with recurrent glioblastoma multiforme (GBM) who require reoperation.
  Interventions: Drug: MK-2206
- Part 2 (Experimental): Participants with GBM and with anaplastic glioma
  Interventions: Drug: MK-2206

INTERVENTIONS:
Drug: MK-2206 — Taken orally once a week

SUMMARY:
MK-2206 is a newly discovered drug that may slow or stop cancer growth. This drug has been used in other research studies, and information from those other research studies suggests that MK-2206 may help to slow or stop the growth of malignant gliomas. In addition, MK-2206 has the capacity to cross the blood-brain barrier. The blood-brain barrier (BBB) is a separation of circulating blood and cerebrospinal fluid (CSF) in the central nervous system (CNS); and although it serves as a protective barrier, it can often interfere with potentially beneficial treatments reaching the brain successfully. Therefore, the investigators hope that because MK-2206 can successfully cross the blood-brain barrier, it will be more effective in patients. The purpose of this study is to see how well MK-2206 works in patients with malignant gliomas and will be conducted in two parts: Part 1 and Part 2.

Part 1 of the study will investigate the effects of MK-2206 on Akt signaling in tumor tissue. Ten patients with recurrent GBM who require reoperation will receive a short pre-operative course of MK-2206. After recovery from surgery, patients will resume MK-2206 until disease progression or the development of unacceptable toxicities. Part 2 of this trial will be initiated only AFTER analysis of Part 1 data shows drug penetration into tumor tissue; if there is no significant drug penetration into the tumor and/or there is no reduction of pAkt levels, progression to Part 2 of the trial will be halted. The primary goal of Part 2 is to determine the therapeutic efficacy of MK-2206 as measured by 6-month progression-free survival (PFS6). In Part 2, 40 participants with GBM and 18 with anaplastic glioma will be treated with MK-2206 weekly at a dose selected on the basis of an ongoing phase 1 study. Treatment duration will be measured in 4-week cycles. Participants will remain on treatment until tumor progression, as long as there are no unacceptable toxicities. Responses will be assessed by clinical examinations every 4 weeks and MRI scans every 8 weeks.

DETAILED DESCRIPTION:
* Participants will have the following tests and procedures within 2 days before the first dose of MK-2206: medical history, physical examination, blood tests, urine tests and EKG.
* Participants in Part 2 of this research study may also have optional FDG-PET imaging done. If the participant agrees, they will have two PET scans performed; one within a week before beginning study drug, and another within 3 days after starting study drug.
* Participants in Part 1 will take MK-2206 orally prior to surgery on days 1-8 (with surgery after the MK-2206 dose on day 8). They will have an EKG within 4-8 hours after their first dose of MK-2206, and again on Day 8. During surgery, a sample of the tumor will be taken for research. The tumor tissue will be analyzed to measure the level of MK-2206 in the tumor and to study the effect of the drug on the tumor. Genetic tests will be done on the tumor tissue to determine if the tumor's genetic profile can predict response to treatment. You will also have 3 teaspoons of blood drawn to measure the level of MK-2206 in the blood. An assessment of the participant's tumor by MRI or CT scan will be done within 96 hours of surgery to determine how much of the tumor has been removed. One to 4 weeks after surgery (within 14 days of the last MRI/CT scan), MK-2206 treatment will restart at the same schedule as before surgery (weekly dosing). Within 2 days prior to restarting MK-2206 the following tests and procedures must be completed: medical history, physical examination, blood tests, urine test and EKG.
* Participants in both groups will receive MK-2206 by mouth once a week (Days 1, 8, 15, and 22). Participants will receive an EKG within 4-8 hours after their first dose of MK-2206 (for Part 1 participants, this is day 1 pre-surgery; for Part 2 participants, this is day 1 of the first cycle of treatment). Participants will receive an EKG weekly during their first cycle of treatment with MK-2206. The following tests and procedures are required within 2 days before the start of each subsequent 4-week cycle of MK-2206 treatment: medical history, physical examination, blood tests, urine test, and EKG. Each treatment cycle lasts 4 weeks during which time participants will be taking the study drug once a week. In addition, patients will also need the following tests/procedures performed during treatment cycles: medical history and physical examination on Day 15 (+/- 2 days) of Cycles 1 and 2 and blood tests weekly during Cycle 1 and on Day 15 (+/- 2 days) of cycle 2.
* Assessments of the tumor by MRI will be performed within one week prior to the start of each odd-numbered cycle, starting with cycle 3.
* Participants can continue to receive study drug until their disease worsens or develop unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioblastoma or gliosarcoma. Participants will be eligible if the orginal histology was low-grade glioma and a subsequent histological diagnosis of glioblastoma or gliosarcoma is made.
* Unequivocal evidence for tumor progression by MRI or CT scan. A scan should be performed within 14 days of registration. The same type of scan must be used throughout the period of protocol treatment for tumor measurement. MRI scans are preferred whenever possible. If participants in Part 2 of the study are taking corticosteroids, the dose must be stable or decreasing for at least 5 days prior to the scan.
* Must have recovered from the toxic effects of prior therapy. From the start of scheduled study treatment, the following time periods must have elapsed: 4 weeks from any investigational agent, 4 weeks from cytotoxic therapy, or 4 weeks from other anti-tumor therapies.
* Must have failed prior radiation therapy and must have an interval of at least 12 weeks from the completion of radiation therapy.
* Prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of progressive disease based upon nuclear imaging, MR spectroscopy, or histopathology.
* Participants having undergone recent resection of recurrent or progressive tumor will be eligible as long as the following conditions apply: a) they have recovered from the effects of surgery, b) residual disease following resection of recurrent tumor is not mandated for eligibility. To best assess the extent of residual disease post-operatively, and MRI or CT scan should be done no later than 96 hours following surgery or at least 4 weeks post-operatively, in either case within 14 days prior to registration. If participants in Part 2 of the study are taking corticosteroids, the dose must be stable or decreasing for at least 5 days prior to the scan. If steroids are added or the steroid dose is increased between the date of the screening MRI or CT scan and the start of treatment, a new baseline MRI or CT is required.
* 18 years of age or older
* Life expectancy of > 8 weeks
* Karnofsky performance status 60 or greater
* Normal organ and marrow function as outlined in the protocol
* At least 35-45 paraffin slides (standard thickness of 4 microns) from any prior surgery available for correlative studies
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.
* Participants must be registered for the Ivy Consortium Tissue and Data Study.

Additional Part 1 Eligibility Criteria:

* Must be deemed by the site Investigator to be an appropriate candidate for surgical resection.
* Must have frozen tumor sample (minimum of 100mg of tissue) from any prior surgery available for correlative studies
* Unequivocal evidence for tumor progression by MRI or CT scan. For this scan only, increasing corticosteroid doses are acceptable.

Additional Part 2 Eligibility Criteria:

* Subjects with anaplastic gliomas who meet other eligibility criteria are eligible.

Exclusion Criteria:

* Participants who have received therapy for more than two prior relapses
* Prior treatment with Akt inhibitors, PI3K inhibitors, mTOR inhibitors, or anti-angiogenic agents
* Must not be on an enzyme-inducing anti-epileptic drug. If previously on an EIAED, the patient must be off of it for at least two weeks prior to registration.
* Receiving any medications or substances that are strong inhibitors or inducers of CYP3A4
* Receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-2206
* History or current evidence of heart disease
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, chronic liver disease, chronic renal disease, chronic pulmonary disease, or psychiatric illness/social situations that would limit compliance with study requirements.
* Poorly controlled diabetes mellitus
* Pregnant or breastfeeding women
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 3 years: cervical cancer in situ, and basal cell squamous cell carcinoma of the skin
* HIV-positive individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Part 1: Akt inhibition | 2 years
  Quantitative pAkt analysis on post-treatment frozen tumor tissue. Equal or more than half of the specimens must demonstrate an absolute pAkt level that is consistent with adequated pAkt inhibition; this threshold has been determined by Merck based on data from prior phase I solid tumor re-biopsy studies.
Part 1: MK-2206 levels in tumor tissue | 2 years
  The level of MK-2206 in tumor tissue.
Part 2: Therapeutic efficacy | 3 years
  Determine the therapeutic efficacy of MK-2206 as measured by progression-free survival at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y. Wen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - UCLA Medical Center, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Memorial Sloan Kettering, New York, New York